CLINICAL TRIAL: NCT05063305
Title: The Efficacy of Probiotics on Immune and Stress Response and Overall Quality of Life
Brief Title: Probiotics, Immunity, Stress, and QofL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: MeriCal LLC (Unknown)
Responsible Party: Principal Investigator, JeJe Noval, Assistant Professor Nutrition and Dietetics, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 5210331
Record Dates: First submitted 2021-09-13; First posted 2021-10-01 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Stress; Quality of Life
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Male Probiotic (Experimental): • Participants will be instructed to take 1 capsule per day for the following 90 days. If a participant misses a day, they should resume taking 1 capsule per day the next day. The capsule should not be crushed or chewed. The capsule may be taken with or without food per participant preference. The participant should consistently take the capsule at a similar time each day (example: always take it in the morning or evening)
  Interventions: Dietary Supplement: Probiotic
- Male Placebo (Placebo Comparator): • Participants will be instructed to take 1 capsule per day for the following 90 days. If a participant misses a day, they should resume taking 1 capsule per day the next day. The capsule should not be crushed or chewed. The capsule may be taken with or without food per participant preference. The participant should consistently take the capsule at a similar time each day (example: always take it in the morning or evening)
  Interventions: Dietary Supplement: Placebo
- Female Probiotic (Experimental): • Participants will be instructed to take 1 capsule per day for the following 90 days. If a participant misses a day, they should resume taking 1 capsule per day the next day. The capsule should not be crushed or chewed. The capsule may be taken with or without food per participant preference. The participant should consistently take the capsule at a similar time each day (example: always take it in the morning or evening)
  Interventions: Dietary Supplement: Probiotic
- Female Placebo (Placebo Comparator): • Participants will be instructed to take 1 capsule per day for the following 90 days. If a participant misses a day, they should resume taking 1 capsule per day the next day. The capsule should not be crushed or chewed. The capsule may be taken with or without food per participant preference. The participant should consistently take the capsule at a similar time each day (example: always take it in the morning or evening)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The probiotic to be used in the study is in capsule form and consists of 12 bacterial strains and 10-billion colony forming unit (CFU). The product consists of the following bacterial strains and species: Bifidobacterium infantis ATCC SD 6720, Bifidobacterium bifidum ATCC SD 6576, Bifidobacterium breve ATCC SD 5206, Bifidobacterium lactis ATCC SD 5220, Bifidobacterium longum ATCC SD 5588, Lactobacillus acidophilus DSM 32754, Lactobacillus casei ATCC SD5213, Lactobacillus paracasei ATCC SD 5275, Lactobacillus plantarum ATCC SD 5209, Lactobacillus reuteri ATCC SD 6689, Lactobacillus rhamnosus ATCC 53103, Lactobacillus salivarius ATCC SD 5208) in combination with the prebiotic, xylooligosacharide (XOS).
  Arms: Female Probiotic; Male Probiotic
Dietary Supplement: Placebo — A placebo, that will be indistinguishable in appearance to the probiotic, will be provided to half of all study participants for the length of the trial. It will contain the following ingredients: Microcrystalline cellulose, magnesium stearate, a vegetarian capsule, and silicon dioxide. The probiotic will be manufactured by MeriCal.
  Arms: Female Placebo; Male Placebo

SUMMARY:
The purpose of this graduate student research study is to evaluate the efficacy of a multi-strain probiotic and investigate if sex differences influence the role of probiotics on stress and immunity biomarkers.

DETAILED DESCRIPTION:
Visit #1

* Participants will read and sign informed consent forms, HIPPA form, and SAHP Covid-19 screening form.
* Participants will perform a baseline oral saliva swab to test for the stress biomarker cortisol and immune markers, including Interleukin-1β (IL-1β) and Tumor Necrosis Factor (TNF).

  * Swabs will be individually packaged. After opening the package, participants will place the swab under their tongue for 1-2 minutes.
  * After swabbing is complete, the swab will be placed into the collection tube and capped immediately.
  * Completed swabs will be placed and held in a sub negative 70° Fahrenheit freezer.
* Participants will complete a Quality-of-Life Questionnaire (10-15 minutes).
* As this study is double blinded, participants will be separated by gender (male and female) and will select a 90-day supply of placebo or probiotic sample at random. For each gender group there will be 50 samples to select from, comprised of a mix of 25 placebo and 25 probiotic bottles.
* Participants will be instructed to take 1 capsule per day for the following 90 days. If a participant misses a day, they should resume taking 1 capsule per day the next day. The capsule should not be crushed or chewed. The capsule may be taken with or without food per participant preference. The participant should consistently take the probiotic at a similar time each day (example: always take it in the morning or evening) Visit #2
* Participants will complete the same Quality-of-Life Questionnaire from visit #1
* Participants will perform a post-study oral saliva swab in the same manner as visit #1

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* 18-90 years of age
* Participants should be of good health

Exclusion Criteria:

* Women who are self-reported as pregnant and/or breastfeeding
* Those who suffer from any systemic illness, such as diabetes mellitus, HIV, cancer, or chronic kidney disease.
* Persons who are diagnosed with clinical depression or anxiety, or other mental health diagnoses such as schizophrenia or Alzheimer's.
* Persons who have taken any probiotic for 5 or more days in the 3 months prior to the trial
* Persons having received antibiotics or non-steroid anti-inflammatory therapy in the last 3-month period prior to the study
* Persons who work night shift
* Persons who consume probiotic rich foods daily, such as yogurt, kimchi, kombucha, kefir, sauerkraut, tempeh, miso, and buttermilk
* Anyone who is allergic to any ingredient in the probiotic or placebo

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Saliva Sample Cortisol | Change in cortisol uL between baseline and 90 days
  Baseline and post-study oral saliva samples will be tested for the stress biomarker cortisol uL.

SECONDARY OUTCOMES:
Saliva Sample IL-1 | Change in Interleukin-1β (IL-1β) uL between baseline and 90 days
  Baseline and post-study oral saliva samples will be tested for Interleukin-1β (IL-1β) uL.
Saliva Sample Tumor Necrosis Factor | Change in Tumor Necrosis Factor (TNF) uL between baseline and 90 days
  Baseline and post-study oral saliva samples will be tested for Tumor Necrosis Factor (TNF) uL.

CONTACTS AND LOCATIONS:
Overall Officials: JeJe Noval, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States